CLINICAL TRIAL: NCT05466045
Title: Using of Extra Virgin Olive Oil in Patient With Hemodialysis to Improve the Effect of Pruritus and Sleep Disorders
Brief Title: Using of Extra Virgin Olive Oil in Hemodialysis Patients to Improve Pruritus and Sleep Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Mei-Hua, Pan, Principal Investigator, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22MMHIS169e
Record Dates: First submitted 2022-07-04; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Uremic Pruritus
Keywords: Pruritus; Hemodialysis; End-stage renal disease (ESRD); Extra virgin olive oil
MeSH Terms: conditions — Pruritus; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Experimental group received olive oil application
  Interventions: Other: Olive oil application in hemodialysis patients with pruritus
- control group (Placebo Comparator): Control group received normal saline application
  Interventions: Other: Normal saline application in hemodialysis patients with pruritus

INTERVENTIONS:
Other: Olive oil application in hemodialysis patients with pruritus — Experimental group: In addition to routine care, a brown glass bottle containing extra virgin olive oil was applied on the itchy skin every 12 hours by rubbing (after washing the patient's face in the morning and after dinner). The intervention duration was 28 days.
  Arms: experimental group
Other: Normal saline application in hemodialysis patients with pruritus — Control group: In addition to routine care, a brown glass bottle containing normal saline was applied on the itchy skin every 12 hours by rubbing (after washing the patient's face in the morning and after dinner). The intervention duration was 28 days.
  Arms: control group

SUMMARY:
Background and Purpose:

Itching is a common complication of hemodialysis patients, which can cause skin damage and affect the patient's comfort. Studies have shown that olive oil is feasible and effective for pain relief, cancer treatment, stroke and cardiovascular disease, as well as wound healing and skin care because it is readily available, natural, and has merely no side effects, and there is no research application on the skin itchiness in hemodialysis patients. The purpose of this study was to investigate the effect of applying extra virgin olive oil to improve skin itching, sleep quality and changes in heart rate variability in hemodialysis patients.

Research method:

This study is designed as a randomized controlled trial (RCT), which is divided into two groups, the experimental group and the control group. Before the interventional measures, a questionnaire pre-test and HRV test are given first, and the interventional measures are given. During the period, in addition to routine care, both groups of patients used a brown roller ball glass bottle containing extra virgin olive oil or normal saline on the itchy skin every 12 hours gently and evenly smeared with fingers , for 28 days, and on the 14th day and 28 days.After intervention, the post-questionnaire test and HRV test were carried out. The research tools include: 5-D 5-D itch scale, Visual Analogue Scale (VAS), Pittsburgh Sleep Quality Index (PSQI) and Heart Rate Variability (HRV) detector.The data collection results were archived with Statistical Package for the Social Sciences (SPSS) statistical software, and the data were processed and analyzed by descriptive statistics, chi-square test, generalized estimating equation (GEE) and independent sample t test.

Expected results: Result showed using extra virgin olive oil can improvement of skin itchiness and sleep quality in hemodialysis patients, and also cost effectiveness of lotions , reduction of drugs burden on kidneys and improvement of patients' quality of life.

DETAILED DESCRIPTION:
Background and Purpose:

Itching is a common complication of hemodialysis patients, which can cause skin damage and affect the patient's comfort. It will not only affect social activities, but also affect the quality of life. In severe cases, it will cause sleep disorders. Studies have shown that olive oil is feasible and effective for pain relief, cancer treatment, stroke and cardiovascular disease, as well as wound healing and skin care because it is readily available, natural, and has no side effects, and there is no research application on the skin itchiness in hemodialysis patients.Therefore the purpose of this study was to investigate the effect of applying extra virgin olive oil to improve skin itching, sleep quality and changes in heart rate variability in hemodialysis patients.

Research method:

This study is designed as a randomized controlled trial (RCT), which is divided into two groups, the experimental group and the control group. The research process is divided into three stages. Before the interventional measures, a questionnaire pre-test and HRV test are given first.The interventional measures are given. During the period, in addition to routine care, both groups of patients used a brown roller ball glass bottle containing extra virgin olive oil or normal saline on the itchy skin every 12 hours gently and evenly smeared with fingers for 28 days. Questionnaire and HRV test were carried on the 14th day .After intervention, the post-questionnaire test and HRV test were carried out. The research tools include: 5-D 5-D itch scale, Visual Analogue Scale (VAS), Pittsburgh Sleep Quality Index (PSQI) and Heart Rate Variability (HRV) detector.The data collection results were archived with Statistical Package for the Social Sciences (SPSS) statistical software, and the data were processed and analyzed by descriptive statistics, chi-square test, generalized estimating equation (GEE) and independent sample t test.

ELIGIBILITY:
Inclusion Criteria:

* ESRD ,Regular hemodialysis patients >3 months

Exclusion Criteria:

* allergic patients
* skin infection
* atopic dermatitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Using of Extra Virgin Olive Oil in Hemodialysis Patients to Improve Pruritus | the 1th ,14th, 28th day
  change of Pruritus
Using of Extra Virgin Olive Oil in Hemodialysis Patients to Improve | the 1th ,14th, 28th day
  change of Sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: mei-hua pan, master, Principal Investigator — Mackay Memorial Hospital

IPD SHARING:
Plan to Share IPD: No